CLINICAL TRIAL: NCT02903290
Title: Longitudinal Monitoring of Energy Expenditure, Dynamic Stability and Fatigue During Gait in Patients With Cerebellar Ataxia Gene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-AOI-10
Record Dates: First submitted 2016-07-22; First posted 2016-09-16 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cerebellar ataxia (Other): Evaluation ataxia according SARAs; measuring the quality of life through SF36 Questionnaire; quantifying the severity of fatigue perceived by FSS questionnaire quantifying the severity of physical tiredness by VAS before and after physical activity; quantified analysis of walking on walking track GAITRite® (with score calculation FAP and GVI) before and after physical activity; physical activity like walking on a treadmill (with measurement of maximal voluntary quadriceps by manual dynamometer before and after physical activity to ensure the induction of fatigue). Patients will be provided with a portable device for analyzing gas exchange FitMateMED® (COSMED, Rome, Italy) during walking analyzes GAITRite®
  Interventions: Other: Longitudinal Monitoring of Energy Expenditure, Dynamic Stability and Fatigue During Gait; Other: walking track GAITRite,manual dynamometer, and treadmill

INTERVENTIONS:
Other: Longitudinal Monitoring of Energy Expenditure, Dynamic Stability and Fatigue During Gait — Longitudinal Monitoring of Energy Expenditure, Dynamic Stability and Fatigue During Gait
Other: walking track GAITRite,manual dynamometer, and treadmill — walking track GAITRite,manual dynamometer, and treadmill

SUMMARY:
Genetic cerebellar ataxias involves progressive degeneration of the cerebellum. Their overall prevalence is estimated at 2-4 cases per 100 000 people. These diseases are manifested by a static and kinetic cerebellar syndrome characterized by impaired balance, coordination, and an ataxic gait. To date, no therapy is available for patients and physical therapy is essential and recommended. The evolution of the pathology causes a degradation of walking, increased instability and risk of falling. In one year, between 74% and 93% of patients reported having fallen at least once. Falls prevention by understanding the mechanisms affecting stability is a major issue in the management of these patients physiotherapy. The analysis of the literature, we assume that there exists a trio "fatigue - instability - energy expenditure" in which the three parameters would influence each other. To date, we do not have data to characterize these interrelationships and their evolution over time.

STUDY OBJECTIVES: The main objective is to study the relationship between changes in energy expenditure and changes in instability when walking at one year in patients with cerebellar ataxia gene. The secondary objectives are to study, after one year of development, the relationship between fatigue, instability, energy consumption, the number of falls, the severity of ataxia and quality of life.

CONDUCT OF THE STUDY: This is a pilot, multicenter, interventional. The projected duration of patient recruitment will be 12 months and the total number of patients will be included in 15. The duration of participation in this study is 12 months for each patient. The anticipated duration of the study is 30 months. Development of the study: Patients included will perform two sets (S1 and S2) tests a year apart including the evaluation of ataxia according Scale for the assessment and rating of ataxia (SARA); measuring the quality of life through SF36 (The Short Form (36)) Questionnaire; quantifying the severity of fatigue perceived by FSS questionnaire quantifying the severity of physical tiredness by VAS before and after physical activity; quantified analysis of walking on walking track GAITRite® (with score calculation FAP and GVI) before and after physical activity; physical activity like walking on a treadmill (with measurement of maximal voluntary quadriceps by manual dynamometer before and after physical activity to ensure the induction of fatigue). Patients will be provided with a portable device for analyzing gas exchange FitMateMED® (COSMED, Rome, Italy) during walking analyzes GAITRite®.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 60;
* Patient with cerebellar syndrome genetically determined or evidence of inheritance;
* Patient walking more than 50 meters independently, with or without technical assistance;
* Patient likely to be followed regularly for at least one year;
* Patient has given written informed consent;
* Patient affiliated to Social Security.

Exclusion Criteria:

* Patient with any other injuries not attributable to the pathology and can influence the running tests according to physician judgment;
* Patient with any disease or condition incompatible to the success of the study according to the doctor's judgment;
* Patient not strolling or sauntering only with a third person to help;
* Major person under guardianship;
* People hospitalized without his consent and not protected by law;
* Nobody deprived of liberty;
* Patients speakers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Pre physical activity scores (Gilette Gait Index (GVI)) to pre exercise walking | At one year
  The main objective is to investigate the relationship between changes in energy expenditure and changes in instability when walking at one year in patients with cerebellar ataxia gene.
Oxygen consumption to pre exercise walking | At one year
  The main objective is to investigate the relationship between changes in energy expenditure and changes in instability when walking at one year in patients with cerebellar ataxia gene.
Pre physical activity scores (Functional Ambulation Performance Score (FAPS)) to pre exercise walking | At one year
  The main objective is to investigate the relationship between changes in energy expenditure and changes in instability when walking at one year in patients with cerebellar ataxia gene.

SECONDARY OUTCOMES:
Functional Systems Scores (FSS) score | At one year
  Study, after one year of development, the relationship between fatigue, instability, energy consumption, the number of falls, the severity of ataxia and quality of life.
Visual Analog Scale (VAS) tiredness | At one year
  Study, after one year of development, the relationship between fatigue, instability, energy consumption, the number of falls, the severity of ataxia and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: SACCONI Sabrina, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France